CLINICAL TRIAL: NCT03639831
Title: ACUTE AND CHRONIC EFFECTS OF A PROPRIETARY BOTANICAL EXTRACT ON ANXIETY, PERCEIVED STRESS, MOOD AND CORTISOL SECRETION AND METABOLISM IN HEALTHY ADULTS: RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-BLIND CLINICAL TRIAL
Brief Title: ACUTE AND CHRONIC EFFECTS OF A BOTANICAL EXTRACT ON ANXIETY, PERCEIVED STRESS, MOOD AND CORTISOL IN HEALTHY ADULTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Activ'inside (Industry)
Collaborators: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PTC198-2017
Record Dates: First submitted 2018-07-03; First posted 2018-08-21 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Mood Disorders
Keywords: Mood; Anxiety; Stress; Dietary supplement; Botanical
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Proprietary, standardized botanical extract
  Interventions: Dietary Supplement: Proprietary, standardized botanical extract
- Placebo group (Placebo Comparator): Placebo (maltodextrin)
  Interventions: Dietary Supplement: Placebo (maltodextrin)

INTERVENTIONS:
Dietary Supplement: Proprietary, standardized botanical extract — 2 capsules/ day providing the proprietary botanical extract as unique active ingredient
  Arms: Active group
Dietary Supplement: Placebo (maltodextrin) — 2 capsules/ day providing no active component
  Arms: Placebo group

SUMMARY:
Mood disorders, including depression and anxiety, are one of the main causes of the overall disease burden worldwide.

In recent years, the efficacy of certain botanicals as an alternative solution for depression has been evaluated in a number of clinical trials.

However, only few studies looked at the effects of these botanicals on mood in healthy subjects.

The aim of the proposed randomised, double-blind, placebo-controlled, parallel groups methodology is to assess the acute and chronic effects of daily supplementation with a proprietary and standardized botanical extract in comparison to placebo in healthy adults aged 18-60 years with self-reported low mood.

DETAILED DESCRIPTION:
The chronic effect of the active product on mood, anxiety, perceived stress, quality of life and cortisol secretion & metabolism will be assessed through validated questionnaires and urine collection after 2, 4 and 8 weeks of daily supplementation.

The acute effect of the product will be assessed after a single dose and exposure to an acute psychological stressor. Before, during and after the stressor, saliva samples will be collected and subjective levels of anxiety and mood will be measured. In addition, Galvanic Skin Response (GSR) and heart rate (HR) will be measured throughout the stressor session.

ELIGIBILITY:
Inclusion Criteria:

* With non-pathological feelings of anxiety and/ or stress in daily life:

  * Subjects self-reporting low mood;
  * Total score ≥ 40 at the Profile of Mood State (POMS 2);
  * Score < 16 at the Generalized Anxiety Disorder 7-item (GAD-7) questionnaire
  * Score ≤ 10 at the Patient Health Questionnaire 9-item (PHQ-9)
  * Not meeting the diagnosis criteria for any mental disorder
* Body Mass Index (BMI) in the normal range: 18.5 ≥ BMI ≤ 30 kg/ m2
* For non-menopausal women: using effective contraception/pregnancy is not physiologically possible.
* Subject showing no difficulty for salivary sampling
* Subjects capable of and willing to comply with the protocol and to give their written informed consent

Main Exclusion Criteria:

* Diagnosis of psychological pathology within the previous 3 years
* Diagnosis of cognitive pathology
* Anxiolytic or antidepressant treatment, within the previous 3 months
* Event likely to have impacted the subject's emotional and/ or psychological state within the last 8 weeks or planned during the next 8 weeks
* Menopausal transition
* High blood pressure
* Subjects diagnosed with diabetes, cardiovascular disease, recurrent infectious diseases or chronic inflammatory pathology
* Usual corticoid treatment/ steroidal anti-inflammatory treatment
* Unbalanced thyroid disease
* High physical activity practice
* Tobacco consumption
* Subjects consuming any food supplement
* Excessive alcohol or caffeine use
* Consumption of recreational drugs
* Subject currently participating in other clinical or nutrition intervention studies, or has done in the past 4 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Mood state | Week 8
  Variation of the Profile of mood states (POMS-2) total score: TMD (Total Mood Disturbance score). The POMS-2 is a scale which includes six mood subscales: Anger, Confusion, Depression, Fatigue, Tension, and Vigor. Each subscale is scored between 0 and 100. TMD is determined by summing the Negative Mood State subscores and subtracting the Vigor subscore (unique Positive Mood State subscale). For each subscale except Vigor, a lower subscore indicates a better mood state. For the Vigor subscale, a higher subscore indicates a better mood state. A lower POMS-2 TMD indicates a better mood state.

SECONDARY OUTCOMES:
POMS-2 subscores | week 2, week 4, week 8
  Variation of the POMS-2 subscores: Anger, Confusion, Depression, Fatigue, Tension, and Vigor. Each subscale is scored between 0 and 100. For each subscale except Vigor, a lower subscore indicates a better mood state. For the Vigor subscale, a higher subscore indicates a better mood state.
Anxiety state State-Trait Anxiety Inventory | week 2, week 4, week 8
  Variation of the State-Trait Anxiety Inventory (STAI-State) score. Min score: 20; Max score: 80. Higher score corresponds to a higher level of anxiety.
Anxiety state according to the Hospital Anxiety and Depression Scale | week 2, week 4, week 8
  Variation of the anxiety subscore of the Hospital Anxiety and Depression Scale (HADS-A). Min score: 0; Max score: 21. Higher score corresponds to a higher level of anxiety.
Percentage of responders | week 2, week 4, week 8
  A responder is defined as a participant with a statistically significant reduction of the POMS-2 TMD T-score. A lower POMS-2 TMD indicates a better mood state.
Psychological stress | week 2, week 4, week 8
  Variation of the Perceived Stress Scale (PSS-10) score (min score: 0; max score: 40; a higher score corresponds to a lower psychological stress feeling)
Worry feeling | week 2, week 4, week 8
  Variation of the Penn State Worry Questionnaire score (min score: 16; max score: 80; a higher score corresponds to a higher worry feeling)
Coping response to stress | week 2, week 4, week 8
  Variations of the COPE inventory score (min score: 60; max score: 240). A higher score indicates that the subject uses more coping strategies in response to stress.
Depressive-like state | week 2, week 4, week 8
  Variation of the depression subscore of the HADS (HADS-D). HADS-D score is comprised between 0 and 21. A higher HADS-D score indicates a higher level of depression.
Quality of life score | week 2, week 4, week 8
  Variation of the World Health Organisation Quality of Life questionnaire (WHOQOL-BREF) score, comprised between 16 and 80. Higher score indicates higher quality of life.
Cognitive performances | week 2, week 4, week 8
  Variation of the performance on serial subtractions tasks: total and correct responses at serials 3s, 7s and 17s. For Serial 3s: Participants will be instructed to count backwards in threes from a given number, as quickly and accurately as possible. For Serial 7s: same task as for serial 3s but with the serial subtraction of 7. Serial 17s: same task as for serial 3s but with the serial subtraction of 17.
Cognitive performances | week 2, week 4, week 8
  Variation of the performance on the tracking task : speed and accuracy. In this task participants are required to use the mouse to move a cursor to attempt to track an asterisk which follows a random on-screen path. The distance between the target and the cursor is then computed every 100 ms.
Diurnal cortisol secretion | week 2, week 4, week 8
  Variation of cortisone/ cortisol urinary concentrations ratio
Diurnal cortisol metabolism | week 2, week 4, week 8
  Variation of allo-tetrahydrocortisol (THFs)/ tetrahydrocortisone (THE) urinary concentrations ratio
Biological response to an acute stressor | week 2, week 4 & week 8; at 15, 30, 45, 60 & 75 min after exposure to the stressor
  Incremental area under the curve (iAUC) of the salivary cortisol concentration and alpha-amylase activity
Psychological response to an acute stressor assessed through the STAI | week 2, week 4 & week 8; 30 and 60 min after exposure to the stressor
  Variation of the State-Trait Anxiety Inventory (STAI-State) score. Min score: 20; Max score: 80. Higher score corresponds to a higher level of anxiety.
Psychological response to an acute stressor assessed on a Visual Analogical Scale | week 2, week 4 & week 8; 30 and 60 min after exposure to the stressor
  Variation of the perceived stress scores obtained at a Visual Analogical Scale (VAS). Score range: 0-100. Higher score indicates a higher level of anxiety.
Hemodynamic response to an acute stressor | week 2, week 4 & week 8; 0 to 15 min after exposure to the stressor
  Maximum increase and incremental area under the curve (iAUC) of the heart rate
Galvanic Skin Response to the acute stressor | week 2, week 4 & week 8
  Averaged raw score in microSiemens (µS) during exposure to acute stressor, likely to be comprised between 0.5 µS and 5 µS. A higher GSR indicates a higher stress state.

OTHER OUTCOMES:
Bioavaialability | week 2, week 4 & week 8
  Urinary metabolites
Biomarqueurs of oxidative damage | week 2, week 4 & week 8
  Change in urine F2-isoprostane

CONTACTS AND LOCATIONS:
Overall Officials: David KENNEDY, PhD, Principal Investigator — Brain, Performance and Nutrition Research Centre - Northumbria University
Locations (1):
- Brain, Performance and Nutrition Research Centre, Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson PA, Forster J, Khan J, Pouchieu C, Dubreuil S, Gaudout D, Moras B, Pourtau L, Joffre F, Vaysse C, Bertrand K, Abrous H, Vauzour D, Brossaud J, Corcuff JB, Capuron L, Kennedy DO. Effects of Saffron Extract Supplementation on Mood, Well-Being, and Response to a Psychosocial Stressor in Healthy Adults: A Randomized, Double-Blind, Parallel Group, Clinical Trial. Front Nutr. 2021 Feb 1;7:606124. doi: 10.3389/fnut.2020.606124. eCollection 2020. PMID 33598475